CLINICAL TRIAL: NCT00973973
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of NBI-56418 Sodium in Subjects With Endometriosis
Brief Title: Efficacy and Safety Study of Elagolix in Women With Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-56418-0901
Record Dates: First submitted 2009-09-07; First posted 2009-09-09 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-04

CONDITIONS: Endometriosis, Pain
Keywords: Pelvic Pain,NBI-56418,Endometriosis
MeSH Terms: conditions — Endometriosis; Pain | interventions — elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elagolix 150 mg (Experimental): Participants received 150 mg elagolix orally once a day for 8 weeks during the double-blind treatment period and continued to receive 150 mg elagolix for 16 additional weeks during the open-label treatment period.
  Interventions: Drug: Elagolix
- Placebo (Placebo Comparator): Participants received placebo orally once a day for 8 weeks during the double-blind treatment period and switched to receive 150 mg elagolix for 16 weeks during the open-label treatment period.
  Interventions: Drug: Placebo; Drug: Elagolix

INTERVENTIONS:
Drug: Placebo — Matching placebo tablets taken orally once a day
  Arms: Placebo
Drug: Elagolix — Immediate release (IR) tablets taken orally once a day
  Other Names: NBI-56418; Orilissa™

SUMMARY:
The purpose of this study is to evaluate elagolix (NBI-56418) compared to placebo for its effects on endometriosis related pelvic pain and its safety.

DETAILED DESCRIPTION:
Participants were randomized (1:1) to 150 mg elagolix once daily or placebo once daily for the first 8 weeks of the study. Following 8 weeks of dosing, participants continued in the study for an additional 16 weeks in an open-label phase where all participants still enrolled in the study received 150 mg elagolix once daily.

There was no pre-specified primary efficacy end point for this study as there is no single key efficacy outcome measure in this exploratory Phase 2 study. However, the efficacy measures of primary interest included the daily assessment of dysmenorrhea, non-menstrual pelvic pain and dyspareunia on a 4-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe) using an e-Diary.

ELIGIBILITY:
Inclusion Criteria:

* Be female, aged 18 to 49 years, inclusive.
* Have moderate to severe pelvic pain due to endometriosis.
* Have a history of regular menstrual cycles.
* Have been surgically (laparoscopy or laparotomy) diagnosed with endometriosis within 8 years of the start of screening.
* Have a Body Mass Index (BMI) of 18 to 36 kg/m², inclusive.
* Agree to use two forms of non-hormonal contraception during the study.

Exclusion Criteria:

* Are currently receiving gonadotropin-releasing hormone (GnRH) agonist, a GnRH antagonist other than NBI-56418, or danazol or have received any of these agents within 6 months of the start of screening.
* Are currently receiving subcutaneous medroxyprogesterone acetate (DMPA-SC) or intramuscular medroxyprogesterone acetate (DMPA-IM) or have received any of these agents within 3 months of the start of screening.
* Are currently using hormonal contraception or other forms of hormonal therapy or received such treatment within the last month.
* Have had surgery for endometriosis within the last month.
* Have had a hysterectomy or bilateral oophorectomy.
* Are using systemic steroids on a chronic or regular basis within 3 months.
* Have uterine fibroids ≥ 3 cm in diameter.
* Have pelvic pain that is not caused by endometriosis.
* Have unstable medical condition or chronic disease.
* Have been pregnant within the last six months.
* Currently breast feeding.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2009-10-12 (Actual); Primary Completion 2010-09-22 (Actual); Study Completion 2010-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 37 centers in the United States.
Pre-assignment Details: The study consisted of up to 8 weeks of screening with data collection to establish baseline pain, an 8-week double-blind placebo-controlled treatment period, a 16-week open-label treatment period with all patients receiving elagolix 150 mg once per day, and a 6-week posttreatment follow-up period.
Period: Double-blind Treatment Phase (Weeks 1-8)
Arm/Group | Placebo | Elagolix 150 mg
Started | 69 | 68
Received Study Drug | 69 | 68
Completed | 63 | 60
Not Completed | 6 | 8
Not completed — Adverse Event | 1 | 3
Not completed — Protocol Deviation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Sponsor/Investigator Decision | 1 | 1
Period: Open-label Treatment Phase (Weeks 8-24)
Arm/Group | Placebo | Elagolix 150 mg
Started | 63 | 60
Completed | 57 | 55
Not Completed | 6 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Deviation | 1 | 0
Not completed — Noncompliance | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Sponsor/Investigator Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Elagolix 150 mg | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (0.9) | 32.8 (0.7) | 32.9 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 68 | 137
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Black | 7 | 6 | 13
  White | 57 | 55 | 112
  Hispanic | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Monthly Mean Dysmenorrhea Score During the Double-blind Treatment Phase
Description: Participants assessed dysmenorrhea (pain during menstruation) and its impact on their daily activities at approximately the same time each day of their period in an electronic diary (e-Diary) according to the following response options:
  * 0 = No discomfort
  * 1 = Mild discomfort but I was easily able to do the things I usually do
  * 2 = Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3 = Severe pain that made it difficult to do the things I usually do.
  The monthly mean dysmenorrhea score is the average of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and Weeks 4 and 8
Population: All randomized participants who received at least 1 dose of study drug and had at least 10 evaluable e-Diary reports during the double-blind period (intent-to-treat population). The analysis includes participants with non-missing data at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 66 | 66
units on a scale
  Week 4 | -0.24 (0.076) | -0.49 (0.076)
  Week 8: number analyzed (Participants) | 64 | 64
  Week 8 | -0.37 (0.107) | -1.13 (0.107)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Comparison of Change from Baseline at Week 4; Test type: Superiority; p = 0.0262, ANCOVA; Analysis of covariance (ANCOVA) model including baseline value as a covariate; LS Mean Difference = -0.24, 95% CI 2-sided [-0.45 to -0.03], Standard Error of Mean 0.107
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 8; Test type: Superiority; p < 0.0001, ANCOVA; Analysis of covariance (ANCOVA) model, including baseline value as a covariate; LS Mean Difference = -0.76, 95% CI 2-sided [-1.06 to -0.46], Standard Error of Mean 0.152

2. Primary Outcome: Change From Baseline in the Monthly Mean Dysmenorrhea Score During the Open-label and Posttreatment Phases
Description: Participants assessed dysmenorrhea (pain during menstruation) and its impact on their daily activities at approximately the same time each day of their period in an electronic diary (e-Diary) according to the following response options:
  * 0 = No discomfort
  * 1 = Mild discomfort but I was easily able to do the things I usually do
  * 2 = Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3 = Severe pain that made it difficult to do the things I usually do.
  The monthly mean dysmenorrhea score is the average of the daily values reported during the 4 weeks prior to each visit, except for the week 30 value which is based on 6 weeks of data.
Time Frame: Baseline and Weeks 12, 16, 20, 24, and 30 (6 weeks posttreatment)
Population: All randomized participants who received at least 1 dose of study drug and had at least 10 evaluable e-Diary reports during the double-blind period (intent-to-treat population) with data on or after Week 12. The analysis includes participants with non-missing data at each time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 61 | 60
units on a scale
  Week 12 | -0.768 (0.118) | -1.060 (0.130)
  Week 16: number analyzed (Participants) | 61 | 59
  Week 16 | -1.325 (0.112) | -1.022 (0.137)
  Week 20: number analyzed (Participants) | 57 | 57
  Week 20 | -1.026 (0.119) | -0.991 (0.121)
  Week 24: number analyzed (Participants) | 57 | 57
  Week 24 | -1.282 (0.118) | -1.372 (0.132)
  Week 30: number analyzed (Participants) | 55 | 55
  Week 30 | -0.547 (0.104) | -0.534 (0.102)

3. Primary Outcome: Change From Baseline in the Monthly Mean Non-menstrual Pelvic Pain Score During the Double-Blind Treatment Phase
Description: Participants assessed their pelvic pain not related to menses and its impact on their daily activities at approximately the same time each day they were not having their period in an e-Diary according to the following response options:
  * 0 = No discomfort
  * 1 = Mild discomfort but I was easily able to do the things I usually do
  * 2 = Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3 = Severe pain that made it difficult to do the things I usually do.
  The monthly mean non-menstrual pelvic pain score is the average of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and weeks 4 and 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 66 | 66
units on a scale
  Week 4 | -0.05 (0.061) | -0.26 (0.061)
  Week 8: number analyzed (Participants) | 64 | 64
  Week 8 | -0.19 (0.071) | -0.47 (0.071)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 4; Test type: Superiority; p = 0.0163, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -0.21, 95% CI 2-sided [-0.38 to -0.04], Standard Error of Mean 0.086
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 8; Test type: Superiority; p = 0.0066, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -0.28, 95% CI 2-sided [-0.48 to -0.08], Standard Error of Mean 0.101

4. Primary Outcome: Change From Baseline in the Monthly Mean Non-menstrual Pelvic Pain Score During the Open-label and Posttreatment Phases
Description: Participants assessed their pelvic pain not related to menses and its impact on their daily activities at approximately the same time each day they were not having their period in an e-Diary according to the following response options:
  * 0 = No discomfort
  * 1 = Mild discomfort but I was easily able to do the things I usually do
  * 2 = Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3 = Severe pain that made it difficult to do the things I usually do.
  The monthly mean non-menstrual pelvic pain score is the average of the daily values reported during the 4 weeks prior to each visit, except for the week 30 value which is based on 6 weeks of data.
Time Frame: Baseline and Weeks 12, 16, 20, 24, and 30 (6 weeks posttreatment)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 61 | 60
units on a scale
  Week 12 | -0.355 (0.087) | -0.727 (0.072)
  Week 16: number analyzed (Participants) | 61 | 59
  Week 16 | -0.422 (0.078) | -0.763 (0.079)
  Week 20: number analyzed (Participants) | 57 | 57
  Week 20 | -0.524 (0.090) | -0.759 (0.082)
  Week 24: number analyzed (Participants) | 57 | 57
  Week 24 | -0.543 (0.092) | -0.801 (0.082)
  Week 30: number analyzed (Participants) | 55 | 55
  Week 30 | -0.326 (0.104) | -0.689 (0.085)

5. Primary Outcome: Change From Baseline in the Monthly Mean Cumulative Pain Score During the Double-Blind Treatment Phase
Description: Participants assessed dysmenorrhea or non-menstrual pelvic pain at approximately the same time each day in an e-Diary according to the following:
  * 0 = No discomfort
  * 1 = Mild discomfort but I was easily able to do the things I usually do
  * 2 = Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3 = Severe pain that made it difficult to do the things I usually do.
  The monthly mean cumulative pain score is the average of the daily values for all days (menstrual and non-menstrual) reported during the 4 weeks prior to each visit.
Time Frame: Baseline and weeks 4 and 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 66 | 66
units on a scale
  Week 4 | -0.11 (0.058) | -0.32 (0.058)
  Week 8: number analyzed (Participants) | 64 | 64
  Week 8 | -0.21 (0.070) | -0.55 (0.070)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 4; Test type: Superiority; p = 0.0089, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -0.22, 95% CI 2-sided [-0.38 to -0.06], Standard Error of Mean 0.082
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 8; Test type: Superiority; p = 0.0011, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -0.33, 95% CI 2-sided [-0.53 to -0.14], Standard Error of Mean 0.100

6. Primary Outcome: Change From Baseline in the Monthly Mean Cumulative Pain Score During the Open-label and Posttreatment Phases
Description: Participants assessed dysmenorrhea or non-menstrual pelvic pain at approximately the same time each day in an e-Diary according to the following:
  * 0: No discomfort
  * 1: Mild discomfort, I was easily able to do the things I usually do
  * 2: Moderate discomfort or pain making it difficult to do some of the things I usually do
  * 3: Severe pain making it difficult to do the things I usually do
  The monthly mean cumulative pain score is the average of the daily values for all days (menstrual and non-menstrual) reported during the 4 weeks prior to each visit, except for the week 30 value which is based on 6 weeks of data.
Time Frame: Baseline and Weeks 12, 16, 20, 24, and 30 (6 weeks posttreatment)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 61 | 60
units on a scale
  Week 12 | -0.433 (0.082) | -0.781 (0.070)
  Week 16: number analyzed (Participants) | 61 | 59
  Week 16 | -0.530 (0.072) | -0.793 (0.083)
  Week 20: number analyzed (Participants) | 57 | 57
  Week 20 | -0.615 (0.085) | -0.798 (0.081)
  Week 24: number analyzed (Participants) | 57 | 57
  Week 24 | -0.655 (0.088) | -0.878 (0.082)
  Week 30: number analyzed (Participants) | 55 | 55
  Week 30 | -0.374 (0.095) | -0.666 (0.085)

7. Primary Outcome: Change From Baseline in the Monthly Mean Dyspareunia Score During the Double-Blind Treatment Phase
Description: Participants assessed their dyspareunia (pain during sexual intercourse) at approximately the same time every day in an e-Diary according to the following response options:
  * 0 = Absent; No discomfort during sexual intercourse
  * 1 = Mild; I was able to tolerate the discomfort during sexual intercourse
  * 2 = Moderate; Intercourse was interrupted due to pain
  * 3 = Severe; I avoided intercourse because of pain
  * Does not apply; I was not sexually active for reasons other than my endometriosis or did not have sexual intercourse
  The monthly mean dyspareunia score is the average of the daily values reported during the 4 weeks prior to each visit. Responses of "does not apply" were not included in the calculations.
Time Frame: Baseline and weeks 4 and 8
Population: All randomized participants who received at least 1 dose of study drug and had at least 10 evaluable e-Diary reports during the double-blind period (intent-to-treat population) with non-missing data at each time point. If a participant's responses were all "does not apply" for that month the score was treated as missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 59 | 53
units on a scale
  Week 4: number analyzed (Participants) | 54 | 49
  Week 4 | -0.07 (0.087) | -0.34 (0.091)
  Week 8: number analyzed (Participants) | 51 | 48
  Week 8 | -0.23 (0.095) | -0.61 (0.098)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Comparison of change form baseline at week 4; Test type: Superiority; p = 0.0360, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -0.27, 95% CI 2-sided [-0.52 to -0.02], Standard Error of Mean 0.127
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 8; Test type: Superiority; p = 0.0070, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -0.38, 95% CI 2-sided [-0.65 to -0.11], Standard Error of Mean 0.137

8. Primary Outcome: Change From Baseline in the Monthly Mean Dyspareunia Score During the Open-label and Posttreatment Phases
Description: Participants assessed their dyspareunia (pain during sexual intercourse) at approximately the same time every day in an e-Diary according to the following response options:
  * 0: Absent; No discomfort during sexual intercourse
  * 1: Mild; I was able to tolerate the discomfort during sexual intercourse
  * 2: Moderate; Intercourse was interrupted due to pain
  * 3: Severe; I avoided intercourse because of pain
  * Does not apply; I was not sexually active for reasons other than my endometriosis or did not have sexual intercourse
  The monthly mean dyspareunia score is the average of the daily values reported during the 4 weeks prior to each visit, except for week 30 which is based on 6 weeks of data. Responses of "does not apply" were not included in the calculations.
Time Frame: Baseline and Weeks 12, 16, 20, 24, and 30 (6 weeks posttreatment)
Population: Randomized participants who received at least 1 dose of study drug and had at least 10 evaluable e-Diary reports during the double-blind period (intent-to-treat population) with data on or after Week 12 and non-missing data at each time point. If a participant's responses were all "does not apply" for that month the score was treated as missing.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 53 | 47
units on a scale
  Week 12: number analyzed (Participants) | 49 | 46
  Week 12 | -0.334 (0.125) | -0.696 (0.112)
  Week 16: number analyzed (Participants) | 49 | 43
  Week 16 | -0.453 (0.114) | -0.738 (0.124)
  Week 20: number analyzed (Participants) | 41 | 41
  Week 20 | -0.492 (0.135) | -0.778 (0.121)
  Week 24: number analyzed (Participants) | 40 | 39
  Week 24 | -0.633 (0.155) | -0.789 (0.115)
  Week 30: number analyzed (Participants) | 44 | 40
  Week 30 | -0.300 (0.118) | -0.730 (0.118)

9. Secondary Outcome: Percentage of Participants With a Response in Monthly Mean Dysmenorrhea Score at Week 8
Description: Participants assessed dysmenorrhea (pain during menstruation) and its impact on their daily activities at approximately the same time each day of their period in an e-Diary according to the following response options:
  * 0: No discomfort
  * 1: Mild discomfort but I was easily able to do the things I usually do
  * 2: Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3: Severe pain that made it difficult to do the things I usually do.
  The monthly mean dysmenorrhea score is the average of the daily values reported during the 4 weeks prior to each time point.
  Response was defined as the percentage of participants with a percent decrease from baseline in the week 8 monthly mean score that was greater than or equal to each specified threshold value (10% through 90% in steps of 10%).
Time Frame: Baseline and Week 8
Population: All randomized participants who received at least 1 dose of study drug and had at least 10 evaluable e-Diary reports during the double-blind period (intent-to-treat population) with non-missing data at baseline and week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 64 | 64
percentage of participants
  10% Reduction | 56.3 | 68.8
  20% Reduction | 43.8 | 68.8
  30% Reduction | 32.8 | 62.5
  40% Reduction | 25.0 | 59.4
  50% Reduction | 15.6 | 54.7
  60% Reduction | 9.4 | 51.6
  70% Reduction | 4.7 | 46.9
  80% Reduction | 3.1 | 43.8
  90% Reduction | 3.1 | 43.8

10. Secondary Outcome: Percentage of Participants With a Response in Monthly Mean Non-menstrual Pelvic Pain Score at Week 8
Description: Participants assessed their pelvic pain not related to menses and its impact on their daily activities at approximately the same time each day they were not having their period in an e-Diary according to the following response options:
  * 0 = No discomfort
  * 1 = Mild discomfort but I was easily able to do the things I usually do
  * 2 = Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3 = Severe pain that made it difficult to do the things I usually do.
  The monthly mean non-menstrual pelvic pain score is the average of the daily values reported during the 4 weeks prior to each time point.
  Response is defined as the percentage of participants with a percent decrease from baseline in the week 8 monthly mean score that was greater than or equal to each specified threshold value (10% through 90% in steps of 10%).
Time Frame: Baseline and Week 8
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 64 | 64
percentage of participants
  10% Reduction | 51.6 | 79.7
  20% Reduction | 40.6 | 68.8
  30% Reduction | 32.8 | 62.5
  40% Reduction | 25.0 | 51.6
  50% Reduction | 25.0 | 32.8
  60% Reduction | 20.3 | 26.6
  70% Reduction | 14.1 | 21.9
  80% Reduction | 9.4 | 10.9
  90% Reduction | 4.7 | 7.8

11. Secondary Outcome: Percentage of Participants With a Response in Monthly Mean Cumulative Pain Score at Week 8
Description: Participants assessed dysmenorrhea or non-menstrual pelvic pain at approximately the same time every day in an e-Diary according to the following:
  * 0 = No discomfort
  * 1 = Mild discomfort
  * 2 = Moderate discomfort or pain
  * 3 = Severe pain
  The monthly mean cumulative pain score is the average of the daily values for all days (menstrual and non-menstrual) in the 4 weeks prior to each time point.
  Response is the percentage of participants with a percent decrease from baseline in the week 8 monthly mean score that was greater than or equal to each specified threshold value (10% through 90% in steps of 10%).
Time Frame: Baseline and Week 8
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 64 | 64
percentage of participants
  10% Reduction | 51.6 | 76.6
  20% Reduction | 40.6 | 70.3
  30% Reduction | 37.5 | 59.4
  40% Reduction | 23.4 | 46.9
  50% Reduction | 20.3 | 37.5
  60% Reduction | 15.6 | 26.6
  70% Reduction | 7.8 | 18.8
  80% Reduction | 3.1 | 9.4
  90% Reduction | 0.0 | 9.4

12. Secondary Outcome: Percentage of Participants With a Response in Monthly Mean Dyspareunia Score at Week 8
Description: Participants assessed their dyspareunia (pain during sexual intercourse) at approximately the same time every day in an e-Diary according to the following response options:
  * 0 = Absent; No discomfort during sexual intercourse
  * 1 = Mild; I was able to tolerate the discomfort during sexual intercourse
  * 2 = Moderate; Intercourse was interrupted due to pain
  * 3 = Severe; I avoided intercourse because of pain
  * Does not apply; I was not sexually active for reasons other than my endometriosis or did not have sexual intercourse
  The monthly mean dyspareunia score is the average of the daily values reported during the 4 weeks prior to each time point.
  Response is defined as the percentage of participants with a percent decrease from baseline in the week 8 monthly mean score that was greater than or equal to each specified threshold value (10% through 90% in steps of 10%).
Time Frame: Baseline and Week 8
Population: All randomized participants who received at least 1 dose of study drug and had at least 10 evaluable e-Diary reports during the double-blind period (intent-to-treat population) with non-missing data at baseline and week 8. If a participant's responses were all "does not apply" for that month the score was treated as missing.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 47 | 45
percentage of participants
  10% Reduction | 44.7 | 73.3
  20% Reduction | 38.3 | 64.4
  30% Reduction | 34.0 | 57.8
  40% Reduction | 27.7 | 53.3
  50% Reduction | 23.4 | 48.9
  60% Reduction | 19.1 | 37.8
  70% Reduction | 19.1 | 31.1
  80% Reduction | 17.0 | 22.2
  90% Reduction | 12.8 | 20.0

13. Secondary Outcome: Change From Baseline in the Percentage of Days of Any Analgesic Use During the Double-Blind Treatment Phase
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of any analgesic use is defined as the number of days in the 4 weeks prior to each study visit that the participant reported the use of an analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline and Weeks 4 and 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 66 | 66
percentage of days
  Week 4 | -5.78 (2.782) | -15.62 (2.782)
  Week 8: number analyzed (Participants) | 64 | 64
  Week 8 | -9.19 (2.763) | -21.63 (2.763)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 4; Test type: Superiority; p = 0.0137, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -9.84, 95% CI 2-sided [-17.63 to -2.05], Standard Error of Mean 3.939
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 8; Test type: Superiority; p = 0.0019, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -12.44, 95% CI 2-sided [-20.19 to -4.70], Standard Error of Mean 3.913

14. Secondary Outcome: Change From Baseline in the Percentage of Days of Any Analgesic Use During the Open-Label and Posttreatment Phases
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of any analgesic use is defined as the number of days in the 4 weeks prior to each study visit (except for week 30 which is based on 6 weeks of data) that the participant reported the use of an analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline and Weeks 12, 16, 20, 24, and 30 (6 weeks posttreatment)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 61 | 60
percentage of days
  Week 12 | -14.91 (3.76) | -27.70 (3.49)
  Week 16: number analyzed (Participants) | 61 | 59
  Week 16 | -18.34 (3.33) | -26.27 (3.71)
  Week 20: number analyzed (Participants) | 57 | 57
  Week 20 | -19.82 (4.05) | -26.35 (4.27)
  Week 24: number analyzed (Participants) | 57 | 57
  Week 24 | -20.63 (4.17) | -29.21 (4.23)
  Week 30: number analyzed (Participants) | 55 | 55
  Week 30 | -11.64 (4.18) | -21.83 (4.30)

15. Secondary Outcome: Change From Baseline in the Percentage of Days of Prescription Analgesic Use During the Double-Blind Treatment Phase
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of prescription analgesic use is defined as the number of days in the 4 weeks prior to each study visit that the participant reported the use of a prescription analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline and Weeks 4 and 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 66 | 66
percentage of days
  Week 4 | 0.92 (1.929) | -5.29 (1.929)
  Week 8: number analyzed (Participants) | 64 | 64
  Week 8 | -0.82 (1.802) | -7.16 (1.802)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 4; Test type: Superiority; p = 0.0244, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -6.21, 95% CI 2-sided [-11.61 to -0.81], Standard Error of Mean 2.728
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 8; Test type: Superiority; p = 0.0141, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -6.35, 95% CI 2-sided [-11.39 to -1.30], Standard Error of Mean 2.549

16. Secondary Outcome: Change From Baseline in the Percentage of Days of Prescription Analgesic Use During the Open-Label and Posttreatment Phases
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of prescription analgesic use is defined as the number of days in the 4 weeks prior to each study visit (except for week 30 which is based on 6 weeks of data) that the participant reported the use of a prescription analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline and Weeks 12, 16, 20, 24, and 30 (6 weeks posttreatment)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 61 | 60
percentage of days
  Week 12 | -2.34 (2.70) | -8.53 (1.66)
  Week 16: number analyzed (Participants) | 61 | 59
  Week 16 | -5.52 (2.26) | -7.52 (1.67)
  Week 20: number analyzed (Participants) | 57 | 57
  Week 20 | -5.21 (2.78) | -6.06 (2.31)
  Week 24: number analyzed (Participants) | 57 | 57
  Week 24 | -5.89 (2.56) | -7.83 (1.89)
  Week 30: number analyzed (Participants) | 55 | 55
  Week 30 | -0.72 (3.07) | -6.06 (2.26)

17. Secondary Outcome: Change From Baseline in the Percentage of Days of Narcotic Analgesic Use During the Double-Blind Treatment Phase
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of narcotic analgesic use is defined as the number of days in the 4 weeks prior to each study visit that the participant reported the use of a narcotic analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline and Weeks 4 and 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 66 | 66
percentage of days
  Week 4 | -0.51 (1.287) | -3.63 (1.287)
  Week 8: number analyzed (Participants) | 64 | 64
  Week 8 | -1.19 (1.369) | -4.71 (1.369)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 4; Test type: Superiority; p = 0.0893, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -3.12, 95% CI 2-sided [-6.72 to 0.49], Standard Error of Mean 1.821
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline at week 8; Test type: Superiority; p = 0.0720, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -3.52, 95% CI 2-sided [-7.35 to 0.32], Standard Error of Mean 1.938

18. Secondary Outcome: Change From Baseline in the Percentage of Days of Narcotic Analgesic Use During the Open-Label and Posttreatment Phases
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of narcotic analgesic use is defined as the number of days in the 4 weeks prior to each study visit (except for week 30 which is based on 6 weeks of data) that the participant reported the use of a narcotic analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline and Weeks 12, 16, 20, 24, and 30 (6 weeks posttreatment)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 61 | 60
percentage of days
  Week 12 | -1.91 (2.16) | -4.79 (1.25)
  Week 16: number analyzed (Participants) | 61 | 59
  Week 16 | -4.03 (1.76) | -3.64 (1.27)
  Week 20: number analyzed (Participants) | 57 | 57
  Week 20 | -2.79 (2.24) | -5.41 (1.64)
  Week 24: number analyzed (Participants) | 57 | 57
  Week 24 | -3.12 (2.20) | -3.92 (1.68)
  Week 30: number analyzed (Participants) | 55 | 55
  Week 30 | 0.75 (2.73) | -3.56 (1.69)

19. Secondary Outcome: Change From Baseline to the End of the Double-blind Treatment Phase in Composite Pelvic Signs and Symptoms Score (CPSSS) Total Score and Component Scores
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration. Each component was scored on a scale of 0 to 3 (0 = absent, 1 = mild, 2 = moderate, and 3 = severe).
  Dysmenorrhea, dyspareunia, and non-menstrual pelvic pain scores are based on the participant's assessment of symptoms during the past 28 days; pelvic tenderness and induration were assessed by the investigator based on findings associated with a pelvic examination.
  The total CPSSS has a maximum possible value of 15 (total score range: 0 to 15, where a lower score indicates less signs and symptoms of endometriosis or better functioning). Individual component scores range from 0 (absent) to 3 (severe).
Time Frame: Baseline and Week 8
Population: All randomized participants who received at least 1 dose of study drug and had at least 10 evaluable e-Diary reports during the double-blind period (intent-to-treat population). The analysis includes participants with non-missing data at baseline and week 8.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 66 | 66
units on a scale
  Total Score: number analyzed (Participants) | 62 | 63
  Total Score | -2.19 (0.359) | -4.45 (0.356)
  Dysmenorrhea Component: number analyzed (Participants) | 63 | 63
  Dysmenorrhea Component | -0.39 (0.127) | -1.44 (0.127)
  Non-menstrual Pelvic Pain Component: number analyzed (Participants) | 63 | 63
  Non-menstrual Pelvic Pain Component | -0.54 (0.101) | -0.90 (0.101)
  Dyspareunia Component: number analyzed (Participants) | 50 | 51
  Dyspareunia Component | -0.46 (0.123) | -0.74 (0.121)
  Pelvic Tenderness Component: number analyzed (Participants) | 62 | 63
  Pelvic Tenderness Component | -0.41 (0.102) | -0.80 (0.101)
  Pelvic Induration Component: number analyzed (Participants) | 62 | 63
  Pelvic Induration Component | -0.38 (0.089) | -0.66 (0.088)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Comparison of the change from baseline in CPSSS total score; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -2.26, 95% CI 2-sided [-3.26 to -1.26], Standard Error of Mean 0.505
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline in CPSSS component of dysmenorrhea score; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -1.05, 95% CI 2-sided [-1.41 to -0.69], Standard Error of Mean 0.180
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline in CPSSS component of non-menstrual pelvic pain score; Test type: Superiority; p = 0.0139, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -0.36, 95% CI 2-sided [-0.64 to -0.07], Standard Error of Mean 0.143
Statistical Analysis 4: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline in CPSSS component of dyspareunia score; Test type: Superiority; p = 0.1052, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -0.28, 95% CI 2-sided [-0.63 to 0.06], Standard Error of Mean 0.173
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline in CPSSS component of pelvic tenderness score; Test type: Superiority; p = 0.0081, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -0.39, 95% CI 2-sided [-0.67 to -0.10], Standard Error of Mean 0.143
Statistical Analysis 6: Comparison: Placebo vs Elagolix 150 mg; Comparison of change from baseline in CPSSS component of induration score; Test type: Superiority; p = 0.0240, ANCOVA; ANCOVA model including baseline value as a covariate; LS Mean Difference = -0.29, 95% CI 2-sided [-0.53 to -0.04], Standard Error of Mean 0.125

20. Secondary Outcome: Change From Baseline to the End of the Open-label Treatment Phase in Composite Pelvic Signs and Symptoms Score (CPSSS) Total Score and Component Scores
Description: as for outcome 19
Time Frame: Baseline and week 24
Population: All randomized participants who received at least 1 dose of study drug and had at least 10 evaluable e-Diary reports during the double-blind period (intent-to-treat population) with data on or after Week 24. The analysis includes participants with non-missing data for each component at baseline and week 24.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 57 | 57
units on a scale
  Total Score: number analyzed (Participants) | 56 | 57
  Total Score | -5.571 (0.451) | -5.404 (0.384)
  Dysmenorrhea Component | -1.544 (0.175) | -1.386 (0.175)
  Non-menstrual Pelvic Pain Component | -1.000 (0.128) | -1.211 (0.127)
  Dyspareunia Component: number analyzed (Participants) | 41 | 43
  Dyspareunia Component | -1.12 (0.17) | -0.77 (0.16)
  Pelvic Tenderness Component: number analyzed (Participants) | 56 | 57
  Pelvic Tenderness Component | -1.000 (0.120) | -1.175 (0.112)
  Pelvic Induration Component: number analyzed (Participants) | 56 | 57
  Pelvic Induration Component | -0.964 (0.142) | -0.807 (0.121)

21. Secondary Outcome: Patient Global Impression of Change During the Double-blind Treatment Phase
Description: The Patient Global Impression of Change (PGIC) is a questionnaire-based assessment of the change in endometriosis pain since the initiation of study drug. The participant was asked to select from one of seven response categories:
  1. Very Much Improved
  2. Much Improved
  3. Minimally Improved
  4. Not Changed
  5. Minimally Worse
  6. Much Worse
  7. Very Much Worse
Time Frame: Weeks 4 and 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 66 | 66
units on a scale
  Week 4: number analyzed (Participants) | 65 | 66
  Week 4 | 3.6 (0.16) | 2.8 (0.16)
  Week 8: number analyzed (Participants) | 63 | 63
  Week 8 | 3.4 (0.18) | 2.4 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Comparison of Patient Global Impression of Change at week 4; Test type: Superiority; p = 0.0012, ANOVA; LS Mean Difference = -0.8, 95% CI 2-sided [-1.2 to -0.3], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg; Comparison of Patient Global Impression of Change at week 8; Test type: Superiority; p = 0.0002, ANOVA; LS Mean Difference = -1.0, 95% CI 2-sided [-1.5 to -0.5], Standard Error of Mean 0.26

22. Secondary Outcome: Patient Global Impression of Change During the Open-Label and Posttreatment Phases
Description: as for outcome 21
Time Frame: Weeks 12, 16, 20, 24, and 30 (6 weeks posttreatment)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 61 | 60
units on a scale
  Week 12: number analyzed (Participants) | 61 | 59
  Week 12 | 2.5 (0.2) | 2.0 (0.1)
  Week 16: number analyzed (Participants) | 60 | 59
  Week 16 | 2.4 (0.2) | 1.8 (0.1)
  Week 20: number analyzed (Participants) | 57 | 57
  Week 20 | 2.2 (0.2) | 2.0 (0.1)
  Week 24: number analyzed (Participants) | 57 | 57
  Week 24 | 2.0 (0.2) | 1.8 (0.1)
  Week 30: number analyzed (Participants) | 55 | 53
  Week 30 | 2.4 (0.2) | 2.2 (0.2)

23. Secondary Outcome: Percentage of Participants With a PGIC Response of Much Improved or Very Much Improved During the Double-blind Treatment Phase
Description: as for outcome 21
Time Frame: Weeks 4 and 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 66 | 66
percentage of participants
  Week 4: number analyzed (Participants) | 65 | 66
  Week 4 | 18.5 [9.0 to 27.9] | 37.9 [26.2 to 49.6]
  Week 8: number analyzed (Participants) | 63 | 63
  Week 8 | 30.2 [18.8 to 41.5] | 60.3 [48.2 to 72.4]
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Comparison of response rates at week 4; Test type: Superiority; p = 0.0136, Pearson chi-squared; Difference = 19.4, 95% CI 2-sided [4.4 to 34.4]
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg; Comparison of response rates at week 8; Test type: Superiority; p = 0.0007, Pearson chi-squared; Difference = 30.2, 95% CI 2-sided [13.6 to 46.7]

24. Secondary Outcome: Percentage of Participants With a PGIC Response of Much Improved or Very Much Improved During the Open-label Treatment Phase
Description: as for outcome 21
Time Frame: Weeks 12, 16, 20, 24, and 30 (6 weeks posttreatment)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 61 | 60
percentage of participants
  Week 12: number analyzed (Participants) | 61 | 59
  Week 12 | 59.0 | 76.3
  Week 16: number analyzed (Participants) | 60 | 59
  Week 16 | 61.7 | 76.3
  Week 20: number analyzed (Participants) | 57 | 57
  Week 20 | 71.9 | 71.9
  Week 24: number analyzed (Participants) | 57 | 57
  Week 24 | 73.7 | 86.0
  Week 30: number analyzed (Participants) | 55 | 53
  Week 30 | 69.1 | 73.6

25. Secondary Outcome: Change From Baseline to the End of the Double-blind Treatment Phase in Endometriosis Health Profile-5 (EHP-5)
Description: The EHP-5 is an instrument to measure health-related quality of life in women with endometriosis. The EHP-5 consists of two parts:
  * A core questionnaire consisting of five questions that measure the impact of endometriosis in areas of pain, control and powerlessness, emotional well-being, social support, and self-image with five response categories for each item (Never, Rarely, Sometimes, Often, Always)
  * A supplemental questionnaire consisting of six additional questions which assess the impact of endometriosis on the areas of work, relationship with children, sexual intercourse, feelings about the medical profession, treatment, and infertility with the same five response categories plus an additional response category of Not Relevant which was not scored.
  The scores associated with each possible outcome category are as follows: never (0), rarely (25), sometimes (50), often (75), and always (100). A negative change from baseline score indicates improvement in quality of life.
Time Frame: Baseline and week 8
Population: All randomized participants who received at least 1 dose of study drug and had at least 10 evaluable e-Diary reports during the double-blind period (intent-to-treat population). The analysis includes participants with non-missing data at baseline and week 8 for each question.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 63 | 63
units on a scale
  Pain | -12.3 (3.2) | -29.0 (3.0)
  Control and Powerlessness | -12.7 (3.2) | -35.3 (3.7)
  Emotional Well-being | -10.3 (2.9) | -17.1 (3.1)
  Social Support | -13.1 (3.5) | -27.8 (3.9)
  Self-image | -7.1 (3.3) | -23.4 (3.5)
  Work: number analyzed (Participants) | 54 | 54
  Work | -13.0 (3.4) | -26.4 (3.4)
  Relationship with Children: number analyzed (Participants) | 25 | 23
  Relationship with Children | -19.0 (4.8) | -31.5 (5.5)
  Sexual Intercourse: number analyzed (Participants) | 56 | 52
  Sexual Intercourse | -14.3 (2.9) | -22.6 (3.8)
  Medical Profession: number analyzed (Participants) | 55 | 50
  Medical Profession | -9.5 (2.9) | -11.5 (3.3)
  Frustration with Treatment: number analyzed (Participants) | 48 | 48
  Frustration with Treatment | -20.8 (5.1) | -36.5 (4.6)
  Concerns with Infertility: number analyzed (Participants) | 47 | 48
  Concerns with Infertility | -10.6 (3.6) | -14.1 (3.3)

26. Secondary Outcome: Change From Baseline to the End of the Open-label Treatment Phase in Endometriosis Health Profile-5 (EHP-5)
Description: The EHP-5 is an instrument to measure health-related quality of life in women with endometriosis. The EHP-5 consists of two parts:
  * A core questionnaire consisting of five questions that measure the impact of endometriosis on areas of pain, control and powerlessness, emotional well-being, social support, and self-image with five response categories for each item (Never, Rarely, Sometimes, Often, Always)
  * A supplemental questionnaire consisting of six additional questions which assess the impact of endometriosis on areas of work, relationship with children, sexual intercourse, feelings about the medical profession, treatment, and infertility with the same five response categories plus an additional response category of Not Relevant which was not scored.
  The scores associated with each possible outcome category are as follows: never (0), rarely (25), sometimes (50), often (75), and always (100). A negative change from baseline score indicates improvement in quality of life.
Time Frame: Baseline and week 24
Population: All randomized participants who received at least 1 dose of study drug and had at least 10 evaluable e-Diary reports during the double-blind period (intent-to-treat population) with data on or after Week 12. The analysis includes participants with non-missing data at baseline and week 24 for each question.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 61 | 60
units on a scale
  Pain: number analyzed (Participants) | 57 | 57
  Pain | -30.3 (3.9) | -36.4 (2.9)
  Control and Powerlessness: number analyzed (Participants) | 57 | 57
  Control and Powerlessness | -35.1 (4.3) | -39.5 (3.5)
  Emotional Well-being: number analyzed (Participants) | 57 | 57
  Emotional Well-being | -22.8 (4.0) | -23.7 (3.3)
  Social Support: number analyzed (Participants) | 57 | 57
  Social Support | -29.8 (4.5) | -37.7 (4.1)
  Self-image: number analyzed (Participants) | 57 | 57
  Self-image | -20.6 (4.3) | -25.9 (3.9)
  Work: number analyzed (Participants) | 48 | 48
  Work | -27.6 (4.4) | -37.0 (3.1)
  Relationship with Children: number analyzed (Participants) | 24 | 20
  Relationship with Children | -39.6 (5.4) | -40.0 (4.2)
  Sexual Intercourse: number analyzed (Participants) | 49 | 46
  Sexual Intercourse | -30.1 (3.9) | -27.2 (4.0)
  Medical Profession: number analyzed (Participants) | 49 | 46
  Medical Profession | -16.8 (4.5) | -19.6 (3.9)
  Frustration with Treatment: number analyzed (Participants) | 43 | 45
  Frustration with Treatment | -40.1 (5.5) | -40.6 (4.4)
  Concerns with Infertility: number analyzed (Participants) | 42 | 45
  Concerns with Infertility | -20.8 (5.0) | -22.8 (3.8)

27. Secondary Outcome: Percentage of Days With Uterine Bleeding During the Double- Blind Treatment Phase
Description: Uterine bleeding was reported daily by participants during the study using the e-Diary.
  The percentage of days a participant reported any bleeding was calculated as the total number of days the participant reported any bleeding ( light, moderate, or heavy) divided by the total number of days the participant had a non-missing e-Diary report of vaginal bleeding in the phase.
Time Frame: Screening (8 weeks prior to day 1) and the double-blind treatment phase (Weeks 1-8)
Population: Participants who received at least one dose of randomized, double-blind study drug (safety analysis set) with non-missing data.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 69 | 68
percentage of days
  Screening | 24.29 (0.96) | 22.98 (1.12)
  Double-Blind Treatment Phase (Weeks 1-8): number analyzed (Participants) | 68 | 67
  Double-Blind Treatment Phase (Weeks 1-8) | 23.91 (1.62) | 14.00 (1.03)

28. Secondary Outcome: Number of Days to First Posttreatment Menses
Description: Defined as the number of days from the last dose of study drug until the start date of the first post-treatment menses.
Time Frame: From last day of study drug up to 6 weeks after the last dose.
Population: Participants who received at least one dose of randomized, double-blind study drug (safety analysis set) with non-missing post-treatment data.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 56 | 58
days | 22.0 [1 to 40] | 25.0 [3 to 45]

ADVERSE EVENTS:
Time Frame: From the first dose of any study drug through week 24. The Placebo treatment group includes data for the 8-week double-blind treatment phase. The Elagolix treatment group included data for the total 24-week treatment period for participants initially randomized to elagolix, and 16-week open-label treatment period for participants initially randomized to placebo.
Groups:
- Placebo: Participants received placebo orally once a day for 8 weeks during the double-blind treatment period.
- Elagolix: Participants initially randomized to elagolix received 150 mg elagolix orally once a day for 8 weeks during the double-blind treatment period and continued to receive 150 mg elagolix for 16 additional weeks during the open-label treatment period.
  Participants originally randomized to placebo were switched to receive 150 mg elagolix for 16 weeks during the open-label treatment period.
Arm/Group | Placebo | Elagolix
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/131
Serious Adverse Events (participants affected / at risk) | 3/69 | 1/131
Other Adverse Events (participants affected / at risk) | 13/69 | 49/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=69) | Elagolix (N=131)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
DEPRESSION SUICIDAL (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=69) | Elagolix (N=131)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 13 (13)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 7 (7)
SINUSITIS (Infections and infestations) | 5 (5) | 8 (9)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 8 (10)
HEADACHE (Nervous system disorders) | 3 (3) | 13 (20)
HOT FLUSH (Vascular disorders) | 1 (1) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.